CLINICAL TRIAL: NCT03390075
Title: Identifying the Effect of Shelf Nutrition Labels on Consumer Purchases, Results of a Natural Experiment and Consumer Survey
Brief Title: The Effect of Shelf Nutrition Labels on Purchases
Status: Completed | Type: Observational
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Chen Zhen, Associate professor of agricultural and applied economics, University of Georgia
Other Study IDs: STUDY00003430
Record Dates: First submitted 2017-11-07; First posted 2018-01-04 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Obesity
Keywords: shelf nutrition label, NuVal
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ResearchNow NuVal shoppers: a convenience sample of 665 shoppers at two NuVal chains.

SUMMARY:
NuVal® shelf nutrition labels rate the nutritional quality of foods on a scale of 1 (worst) to 100 (best). In 2014, NuVal updated their nutrient profiling system which changed the NuVal score on many foods. The investigators took advantage of this "natural experiment" to assess the extent to which a change in the NuVal score at a grocery chain influenced yogurt purchases, a category with a wide range of more and less healthy alternatives. The investigators supplemented the retail scanner data with a survey of consumers in stores using NuVal labels to obtain their experience with the labels and the extent to which they state it influences their purchases.

ELIGIBILITY:
Inclusion Criteria:

* US adults regularly shopping at one of two retail chains using NuVal

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: US grocery shoppers
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2016-06-04 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Diet quality as measured by the NuVal scores of yogurt purchased | From 12/30/12 to 8/22/15
  The investigators measured diet quality using weekly yogurt sales data supplied by a US grocery chain. Using an econometric model of yogurt demand, the investigators associated changes in yogurt sales volume for each product before and after the NuVal score change with the direction and magnitude of the score change.

SECONDARY OUTCOMES:
Knowledge and stated use of NuVal labels by participants of an online survey | June 2016
  The investigators conducted an online survey of 665 adult shoppers of two grocery chains that adopted NuVal. The survey elicited participants' awareness of the label, knowledge of NuVal, and stated use of NuVal and other nutrition labels.

REFERENCES:
- [Derived] Finkelstein EA, Li W, Melo G, Strombotne K, Zhen C. Identifying the effect of shelf nutrition labels on consumer purchases: results of a natural experiment and consumer survey. Am J Clin Nutr. 2018 Apr 1;107(4):647-651. doi: 10.1093/ajcn/nqy014. PMID 29635504